CLINICAL TRIAL: NCT06890884
Title: A Randomized, Open-label, Multicenter, Phase 2 Study Evaluating the Efficacy and Safety of Zilovertamab Vedotin (MK-2140) Plus R-CHP Versus Polatuzumab Vedotin Plus R-CHP in Treatment-naïve Participants With GCB Subtype of Diffuse Large B-cell Lymphoma (DLBCL)
Brief Title: A Clinical Study of Zilovertamab Vedotin (MK-2140) Plus Rituximab Plus Cyclophosphamide, Doxorubicin, and Prednisone (R-CHP) Versus Polatuzumab Vedotin Plus R-CHP in People With Diffuse Large B-cell Lymphoma (DLBCL) (MK-2140-011/waveLINE-011)
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2140-011; 2024-515526-89-00 (Registry Identifier: EU CT); U1111-1309-2852 (Registry Identifier: UTN); MK-2140-011 (Other: MSD); waveLINE-011 (Other: MSD); jRCT2021250001 (Registry Identifier: Japan Registry of Clinical Trials (jRCT))
Record Dates: First submitted 2025-03-20; First posted 2025-03-24 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Lymphoma, Large B-Cell, Diffuse
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse | interventions — Rituximab; Cyclophosphamide; Doxorubicin; Prednisone; Prednisolone; polatuzumab vedotin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Zilovertamab vedotin + Rituximab + Cyclophosphamide, Doxorubicin, Prednisone (R-CHP) (Experimental): Participants will receive a dose of zilovertamab vedotin (1.75 mg/kg) plus 750 mg/m^2 cyclophosphamide, 50 mg/m^2 doxorubicin, and 375 mg/m^2 rituximab or rituximab biosimilar administered by intravenous (IV) infusion on Day 1 of each 3-week cycle for up to 6 cycles (up to approximately 4 months) plus 2 additional cycles of rituximab or biosimilar for participants with high risk DLBCL. Participants will also receive 100 mg prednisone or prednisolone via oral tablet per day during Days 1-5 of each 3-week cycle for up to 6 cycles (up to approximately 4 months).
  Interventions: Biological: Zilovertamab vedotin; Biological: Rituximab; Drug: Cyclophosphamide; Drug: Doxorubicin; Biological: Rituximab Biosimilar; Drug: Prednisone; Drug: Prednisolone; Drug: Rescue Medication
- Polatuzumab vedotin + R-CHP (Active Comparator): Participants will receive a dose of polatuzumab vedotin (1.8 mg/kg) plus 750 mg/m^2 cyclophosphamide, 50 mg/m^2 doxorubicin, and 375 mg/m^2 rituximab or rituximab biosimilar administered by IV infusion on Day 1 of each 3-week cycle for up to 6 cycles (up to approximately 4 months) plus 2 additional cycles of rituximab or biosimilar for participants with high risk DLBCL. Participants will also receive 100 mg prednisone or prednisolone via oral tablet per day during Days 1-5 of each 3-week cycle for up to 6 cycles (up to approximately 4 months).
  Interventions: Biological: Rituximab; Drug: Cyclophosphamide; Drug: Doxorubicin; Biological: Rituximab Biosimilar; Drug: Prednisone; Drug: Prednisolone; Biological: Polatuzumab vedotin; Drug: Rescue Medication

INTERVENTIONS:
Biological: Zilovertamab vedotin — IV infusion
  Other Names: MK-2140; VLS-101
  Arms: Zilovertamab vedotin + Rituximab + Cyclophosphamide, Doxorubicin, Prednisone (R-CHP)
Biological: Rituximab — IV infusion
  Other Names: RITUXAN®
Drug: Cyclophosphamide — IV infusion
  Other Names: CYTOXAN®; NEOSAR®
Drug: Doxorubicin — IV infusion
  Other Names: ADRIAMYCIN®
Biological: Rituximab Biosimilar — IV infusion
  Other Names: TRUXIMA®; RUXIENCE®; RIABNI®
Drug: Prednisone — Oral administration or IV infusion
Drug: Prednisolone — Oral administration or IV infusion
Biological: Polatuzumab vedotin — IV infusion
  Arms: Polatuzumab vedotin + R-CHP
Drug: Rescue Medication — Participants receive rescue medication at the investigators discretion, per approved product label. Recommended rescue medication is Granulocyte Colony-Stimulating Factor (G-CSF).

SUMMARY:
Researchers are looking for ways to treat germinal center B-cell-like diffuse large B-cell lymphoma (GCB DLBCL). DLBCL is a fast-growing blood cancer that affects B-cells. GCB is a type of DLBCL that affects young B-cells that are still maturing.

The goal of this study is to learn if more people who receive zilovertamab vedotin (MK-2140) and R-CHP have the cancer respond (go away) than those who receive polatuzumab vedotin and R-CHP.

ELIGIBILITY:
Inclusion Criteria:

The main inclusion criteria include but are not limited to the following:

* Has histologically confirmed diagnosis of germinal center B-cell (GCB) subtype of diffuse large B-cell lymphoma (DLBCL), by prior biopsy, according to the World Health Organization (WHO) classification of neoplasms of the hematopoietic and lymphoid tissues.
* Has positron emission tomography (PET) positive disease at screening, defined as 4 to 5 on the Lugano 5-point scale.
* Has received no prior treatment for their DLBCL.
* Human immunodeficiency virus (HIV) infected participants must have well controlled HIV on antiretroviral therapy (ART).
* Participants who are hepatitis B surface antigen (HBsAg) positive are eligible if they have received hepatitis B virus (HBV) antiviral therapy and have undetectable HBV viral load prior to randomization.
* Participants with history of hepatitis C virus (HCV) infection are eligible if HCV viral load is undetectable at screening.

Exclusion Criteria:

The main exclusion criteria include but are not limited to the following:

* Has a history of transformation of indolent disease to DLBCL.
* Has received a diagnosis of primary mediastinal B-cell lymphoma (PMBCL) or Grey zone lymphoma.
* Has Ann Arbor Stage I DLBCL.
* Has clinically significant (i.e., active) cardiovascular disease: cerebral vascular accident/stroke (<6 months prior to enrollment), myocardial infarction (<6 months prior to enrollment), unstable angina, congestive heart failure (New York Heart Association Classification Class ≥II), or serious cardiac arrhythmia requiring medication.
* Has clinically significant pericardial or pleural effusion.
* Has ongoing Grade >1 peripheral neuropathy.
* Has a demyelinating form of Charcot-Marie-Tooth disease.
* HIV-infected participants with a history of Kaposi's sarcoma and/or Multicentric Castleman's Disease.
* Has ongoing corticosteroid therapy.
* Known additional malignancy that is progressing or has required active treatment within the past 2 years.
* Known active central nervous system (CNS) lymphoma.
* Has active autoimmune disease that has required systemic treatment in the past 2 years.
* Has active infection requiring systemic therapy.
* Has active HBV (defined as HBsAg positive and detectable HBV deoxyribonucleic acid (DNA)) and HCV (defined as anti-HCV antibody positive and detectable HCV ribonucleic acid (RNA)) infection.
* Has history of stem cell/solid organ transplant.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 594 (Estimated)
Dates: Start 2025-04-11 (Actual); Primary Completion 2027-12-13 (Estimated); Study Completion 2032-12-16 (Estimated)

PRIMARY OUTCOMES:
Complete Response Rate (CRR) at End of Treatment (EOT) per Lugano Response Criteria | Up to approximately 31 months
  CRR at EOT is defined as the percentage of participants who experience complete response (CR) per Lugano response criteria as assessed by blinded independent central review (BICR) at end of treatment. CR is complete metabolic (no/minimal FDG uptake) and radiologic response (target lesions regress to ≤1.5 cm in longest transverse diameter of a lesion) and no new lesions. Participants with missing data or who discontinue treatment or study prior to reaching EOT will be considered non-responders and included in the total number of participants.

SECONDARY OUTCOMES:
Progression-free Survival (PFS) per Lugano Response Criteria | Up to approximately 51 months
  PFS is defined as the time from randomization to the first documented disease progression per Lugano response criteria by BICR or death due to any cause, whichever occurs first.
Overall Survival (OS) | Up to approximately 87 months
  OS is defined as the time from randomization to death due to any cause.
Event-free Survival (EFS) per Lugano Response Criteria | Up to approximately 51 months
  EFS is defined as the time from randomization to any of the following events: progressive disease per Lugano response criteria by BICR, death due to any cause, initiation of a new anti-caner therapy, or a positive biopsy for residual disease. The EFS for all participants will be presented.
Duration of CR | Up to approximately 51 months
  For participants who demonstrate CR at EOT per Lugano response criteria by BICR, duration of complete response is defined as the time from the first documented evidence of CR at or before EOT until disease progression or death due to any cause, whichever occurs first.
Number of participants who experience one or more adverse events (AEs) | Up to approximately 9 months
  An AE is defined as any untoward medical occurrence in a participant, temporally associated with the use of study treatment, whether or not considered related to the study treatment. The number of participants who experience at least one AE will be presented.
Number of participants who discontinue study intervention due to an AE | Up to approximately 6 months
  An AE is defined as any untoward medical occurrence in a participant, temporally associated with the use of study treatment, whether or not considered related to the study treatment. The number of participants who experience at least one AE will be presented.
Change From Baseline in Health-Related Quality Of Life (HRQoL) on Functional Assessment of Cancer Therapy Lymphoma (FACT-Lym) Trial Outcome Index (TOI) | Baseline and up to Week 25
  The FACT-Lym is a 42-item questionnaire designed to measure HRQoL and cancer-specific symptoms in non-Hodgkin lymphoma patients. Subscales include FACT-General (FACT-G), FACT-Trial Outcome Index (FACT-TOI), FACT-Lym total score (FACT-Lym TS), and the Lymphoma subscale (Lym S). The Lym S has a single domain consisting of 15 items specific to lymphoma burden with a score ranging from 0 to 60. FACT-G has 4 well-being domains, physical (7 items), social/family (7), emotional (6), and functional (7), with scores ranging from 0 to 108. FACT-TOI combines FACT-G's physical and functional domains with Lym S, with scores ranging from 0 to 116. FACT-Lym TS combines FACT-G with Lym S, with scores ranging from 0 to 168. The scoring of FACT-Lym is on a 5-point Likert scale from 0 to 4, with 0= not at all, 1= a little bit, 2= somewhat, 3=quite a bit, 4=very much. The higher the score the better the quality of life.
Change From Baseline in HRQoL on FACT-Lym Total Score | Baseline and up to Week 25
  The FACT-Lym is a 42-item questionnaire designed to measure HRQoL and cancer-specific symptoms in non-Hodgkin lymphoma patients. Subscales include FACT-General (FACT-G), FACT-Trial Outcome Index (FACT-TOI), FACT-Lym total score (FACT-Lym TS), and the Lymphoma subscale (Lym S). The Lym S has a single domain consisting of 15 items specific to lymphoma burden with a score ranging from 0 to 60. FACT-G has 4 well-being domains, physical (7 items), social/family (7), emotional (6), and functional (7), with scores ranging from 0 to 108. FACT-TOI combines FACT-G's physical and functional domains with Lym S, with scores ranging from 0 to 116. FACT-Lym TS combines FACT-G with Lym S, with scores ranging from 0 to 168. The scoring of FACT-Lym is on a 5-point Likert scale from 0 to 4, with 0= not at all, 1= a little bit, 2= somewhat, 3=quite a bit, 4=very much. The higher the score the better the quality of life.
Change From Baseline in HRQoL on FACT-Lym Physical Well-being (PWB) (Items General Physical [GP]1 through GP7) | Baseline and up to Week 25
  The FACT-Lym is a 42-item questionnaire designed to measure HRQoL and cancer-specific symptoms in non-Hodgkin lymphoma patients. Subscales include FACT-General (FACT-G), FACT-Trial Outcome Index (FACT-TOI), FACT-Lym total score (FACT-Lym TS), and the Lymphoma subscale (Lym S). The Lym S has a single domain consisting of 15 items specific to lymphoma burden with a score ranging from 0 to 60. FACT-G has 4 well-being domains, physical (7 items), social/family (7), emotional (6), and functional (7), with scores ranging from 0 to 108. FACT-TOI combines FACT-G's physical and functional domains with Lym S, with scores ranging from 0 to 116. FACT-Lym TS combines FACT-G with Lym S, with scores ranging from 0 to 168. The scoring of FACT-Lym is on a 5-point Likert scale from 0 to 4, with 0= not at all, 1= a little bit, 2= somewhat, 3=quite a bit, 4=very much. The higher the score the better the quality of life.
Change From Baseline in HRQoL on Functional Assessment of Cancer Therapy/Gynecologic Oncology Group-Neurotoxicity (FACT/GOG-NTX) Neurotoxicity Subscale Score | Baseline and up to Week 25
  The FACT/GOG-NTX provides a targeted assessment of symptoms of peripheral neuropathy, including sensory, motor, and auditory problems and cold sensitivity. It is an 11-item questionnaire designed to measure the neurotoxicity subscale. The scoring of FACT/GOG-NTX is on a 5-point Likert scale from 0 to 4, with 0= not at all, 1= a little bit, 2= somewhat, 3=quite a bit, 4=very much. To produce a Neurotoxicity Subscale score (range 0-44), the sum of the item scores are multiplied by the number of items in the subscale, then divided by the number of items answered.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (106):
- United States (60):
  - Infirmary Cancer Care ( Site 0157), Mobile, Alabama
  - Palo Verde Cancer Specialists ( Site 0105), Glendale, Arizona
  - Genesis Cancer and Blood Institute ( Site 0193), Hot Springs, Arkansas
  - Roy and Patricia Disney Family Cancer Center - Providence Saint Joseph Medical Center ( Site 0135), Burbank, California
  - Bass Medical Group ( Site 0123), Walnut Creek, California
  - Rocky Mountain Cancer Centers (RMCC) ( Site 8001), Aurora, Colorado
  - Colorado West Healthcare System-Grand Valley Oncology ( Site 0165), Grand Junction, Colorado
  - Medical Oncology Hematology Consultants (MOHC) ( Site 8007), Newark, Delaware
  - Georgetown University Medical Center ( Site 0117), Washington D.C., District of Columbia
  - Boca Raton Regional Hospital-Lynn Cancer Institute ( Site 0130), Boca Raton, Florida
  - Mount Sinai Cancer Center ( Site 0140), Miami Beach, Florida
  - Mid Florida Hematology and Oncology Center ( Site 0152), Orange City, Florida
  - Beacon Cancer Care ( Site 0142), Post Falls, Idaho
  - University of Chicago Medical Center ( Site 0126), Chicago, Illinois
  - Illinois Cancer Care ( Site 7005), Peoria, Illinois
  - University of Iowa-Holden Comprehensive Cancer Center ( Site 0139), Iowa City, Iowa
  - Mission Blood & Cancer Care ( Site 0114), Waukee, Iowa
  - Saint Elizabeth Medical Center Edgewood ( Site 0141), Edgewood, Kentucky
  - Baptist Health Hardin ( Site 0154), Elizabethtown, Kentucky
  - Baptist Health Lexington ( Site 0127), Lexington, Kentucky
  - Norton Women's and Children's Hospital-Norton Cancer Institute - St. Matthews ( Site 0185), Louisville, Kentucky
  - Our Lady of the Lake Physician Group-Medical Oncology ( Site 0180), Baton Rouge, Louisiana
  - Minnesota Oncology Hematology (MNO) ( Site 8004), Burnsville, Minnesota
  - Bozeman Health Deaconess Hospital ( Site 0183), Bozeman, Montana
  - NHO Revive Research Institute, LLC ( Site 0121), Lincoln, Nebraska
  - University Of Nebraska Medical Center ( Site 0110), Omaha, Nebraska
  - Atlantic Health Morristown Medical Center ( Site 0163), Morristown, New Jersey
  - Valley Health Systems - Ridgewood Campus ( Site 0125), Paramus, New Jersey
  - Erie County Medical Center ( Site 0175), Buffalo, New York
  - Roswell Park Cancer Institute ( Site 0192), Buffalo, New York
  - Perlmutter Cancer Center at NYU Langone Hospital - Long Island ( Site 0208), Mineola, New York
  - Laura and Isaac Perlmutter Cancer Center at NYU Langone ( Site 0108), New York, New York
  - SUNY Upstate Cancer Center ( Site 0178), Syracuse, New York
  - Clinical Research Alliance ( Site 0122), Westbury, New York
  - University of North Carolina Medical Center ( Site 0136), Chapel Hill, North Carolina
  - Novant Health Presbyterian Medical Center ( Site 0177), Charlotte, North Carolina
  - Novant Health Forsyth Medical Center ( Site 0206), Winston-Salem, North Carolina
  - University of Cincinnati Medical Center ( Site 0156), Cincinnati, Ohio
  - University Hospitals of Cleveland ( Site 0155), Cleveland, Ohio
  - Fairview Hospital-Moll Cancer Center ( Site 0198), Cleveland, Ohio
  - Cleveland Clinic Main ( Site 0101), Cleveland, Ohio
  - Cleveland Clinic - Hillcrest Hospital-Hillcrest Hospital Cancer Center ( Site 0199), Mayfield Heights, Ohio
  - Providence Portland Medical Center ( Site 0120), Portland, Oregon
  - Providence Oncology and Hematology Clinic Westside ( Site 0179), Portland, Oregon
  - Alliance Cancer Specialists (ACS) ( Site 8010), Horsham, Pennsylvania
  - Cancer Care Associates Of York ( Site 0174), York, Pennsylvania
  - Tennessee Cancer Specialists ( Site 7004), Knoxville, Tennessee
  - SCRI Oncology Partners ( Site 7002), Nashville, Tennessee
  - Texas Oncology - West Texas ( Site 8008), Amarillo, Texas
  - Texas Oncology - Central/South Texas ( Site 8006), Austin, Texas
  - Texas Oncology - Northeast Texas ( Site 8002), Palestine, Texas
  - Texas Oncology - San Antonio ( Site 8009), San Antonio, Texas
  - The University of Texas Health Science Center at Tyler dba UT Health East Texas HOPE Cancer Center ( Site 0145), Tyler, Texas
  - Intermountain Medical Center ( Site 0182), Murray, Utah
  - Intermountain Healthcare - St. George ( Site 0203), St. George, Utah
  - Virginia Cancer Specialists, PC ( Site 8003), Manassas, Virginia
  - VCU Health Adult Outpatient Pavillion ( Site 0138), Richmond, Virginia
  - Northwest Cancer Specialists (Compass Oncology) ( Site 8000), Vancouver, Washington
  - SSM Health Dean Medical Group ( Site 0106), Madison, Wisconsin
  - MEDICAL COLLEGE OF WISCONSIN ( Site 0103), Milwaukee, Wisconsin
- Belgium (5):
  - AZ Sint-Maarten, Campus Leopoldstraat 2 ( Site 0306), Mechelen, Antwerpen
  - Cliniques Universitaires Saint-Luc ( Site 0302), Brussels, Bruxelles-Capitale, Region de
  - Hopital de Jolimont ( Site 0304), Haine-Saint-Paul, Hainaut
  - UZ Leuven ( Site 0301), Leuven, Vlaams-Brabant
  - AZ Delta ( Site 0303), Roeselare, West-Vlaanderen
- Germany (2):
  - Uniklinik Erlangen ( Site 0412), Erlangen, Bavaria
  - Universitaetsklinikum Wuerzburg ( Site 0401), Würzburg, Bavaria
- Ireland (2):
  - Mater Misercordiae University Hospital ( Site 0501), Dublin
  - University Hospital Limerick ( Site 0503), Limerick
- Israel (7):
  - Soroka Medical Center ( Site 0606), Beersheba
  - Rambam Health Care Campus ( Site 0604), Haifa
  - Edith Wolfson Medical Center ( Site 0602), Holon
  - Haddasah Medical Center ( Site 0601), Jerusalem
  - Rabin Medical Center ( Site 0607), Petah Tikva
  - Sheba Medical Center ( Site 0603), Ramat Gan
  - ZIV Medical Center ( Site 0605), Safed
- Italy (7):
  - Azienda Ospedaliero-Universitaria SS. Antonio e Biagio e Cesare Arrigo ( Site 0703), Alessandria, Ancona
  - IRCCS - Istituto Romagnolo per lo Studio dei Tumori (IRST) "Dino Amadori" ( Site 0707), Meldola, Forli-Cesena
  - Istituto Clinico Humanitas ( Site 0704), Rozzano, Milano
  - Istituto Europeo di Oncologia ( Site 0701), Milan
  - Universita degli Studi di Napoli Federico II ( Site 0705), Napoli
  - Az. Osp. Ospedali Riuniti VILLA SOFIA-CERVELLO ( Site 0702), Palermo
  - Arcispedale Santa Maria Nuova ( Site 0706), Reggio Emilia
- Japan (9):
  - Aichi Cancer Center ( Site 1007), Nagoya, Aichi-ken
  - Fujita Health University Hospital ( Site 1003), Toyoake, Aichi-ken
  - Hokkaido University Hospital ( Site 1004), Sapporo, Hokkaido
  - National Hospital Organization Sendai Medical Center ( Site 1005), Sendai, Miyagi
  - Kansai Medical University Hospital ( Site 1006), Hirakata, Osaka
  - Shimane University Hospital ( Site 1002), Izumo, Shimane
  - Nippon Medical School Hospital ( Site 1001), Bunkyo, Tokyo
  - National Cancer Center Hospital ( Site 1009), Chūō, Tokyo
  - Nagasaki University Hospital ( Site 1008), Nagasaki
- Poland (5):
  - Pratia MCM Krakow ( Site 0804), Karkow, Lesser Poland Voivodeship
  - Szpital Specjalistyczny im. Jedrzeja Sniadeckiego w Nowym Saczu ( Site 0806), Nowy Sącz, Lesser Poland Voivodeship
  - Narodowy Instytut Onkologii im. Marii Sklodowskiej-Curie ( Site 0803), Warsaw, Masovian Voivodeship
  - Uniwersyteckie Centrum Kliniczne ( Site 0802), Gdansk, Pomeranian Voivodeship
  - Pratia Onkologia Katowice ( Site 0801), Katowice, Silesian Voivodeship
- United Kingdom (9):
  - Bristol Haematology and Oncology Centre ( Site 0908), Bristol, Bristol, City of
  - Stoke Mandeville Hospital ( Site 0917), Aylesbury, Buckinghamshire
  - Royal Devon & Exeter Hospital ( Site 0910), Exeter, Devon
  - University Hospitals Plymouth NHS Trust ( Site 0905), Plymouth, Devon
  - The James Cook University Hospital ( Site 0909), Middlesbrough, England
  - Lincoln County Hospital ( Site 0906), Lincoln, Lincolnshire
  - Hammersmith Hospital ( Site 0915), London, London, City of
  - Clatterbridge Cancer Centre - Liverpool ( Site 0911), Liverpool
  - Christie Hospital NHS Trust ( Site 0901), Manchester

IPD SHARING:
Plan to Share IPD: Yes
https://trialstransparency.msdclinicaltrials.com/pdf/ProcedureAccessClinicalTrialData.pdf
URL: https://externaldatasharing-msd.com/

REFERENCES:
- See also: Merck Clinical Trials Information — https://www.merckclinicaltrials.com/